CLINICAL TRIAL: NCT01858558
Title: Randomized Phase II Study of Autologous Stem Cell Transplantation With Tadalafil and Lenalidomide Maintenance With or Without Activated Marrow Infiltrating Lymphocytes (MILs) in High Risk Myeloma
Brief Title: Tadalafil and Lenalidomide Maintenance With or Without Activated Marrow Infiltrating Lymphocytes (MILs) in High Risk Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1343; NA_00084466 (Other: JHMIRB)
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aMIL Arm (Experimental): Patients receive activated Marrow Infiltrating Lymphocytes (aMIL)
  Interventions: Biological: aMIL; Drug: No aMIL
- No aMIL (Active Comparator): Patients do not receive activated Marrow Infiltrating Lymphocytes (aMIL)
  Interventions: Drug: No aMIL

INTERVENTIONS:
Biological: aMIL — On day 0, patients will receive auto transplant followed by Tadalafil and aMIL. At day 60, patients will receive Lenalidomide.
  Arms: aMIL Arm
Drug: No aMIL — On day 0, patients will receive auto transplant followed by Tadalafil. At day 60, patients will receive Lenalidomide.

SUMMARY:
This research is being done to find out if altering the immune system by giving activated marrow infiltrating lymphocytes (MILs) can improve outcomes for multiple myeloma patients who receive a standard autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years old;
* Patients with active myeloma requiring systemic treatment;
* Newly diagnosed patients. Relapsed myeloma patients that have not previously had a transplant;
* Meeting criteria for high-risk disease;
* Measurable serum and/or urine M-protein from prior to induction therapy documented and available. A positive serum free lite assay is acceptable;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2 (see Appendix C).
* Meet all institutional requirements for autologous stem cell transplantation;
* The patient must be able to comprehend and have signed the informed consent;
* Patients must have had > than PR after last therapy.

Exclusion Criteria:

* Diagnosis of any of the following cancers:

  * POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein] and skin changes);
  * Non-secretory myeloma (no measurable protein on Serum Free Lite Assay);
  * Plasma cell leukemia;
* Diagnosis of amyloidosis;
* Failed to achieve at least a partial response (PR) to latest therapy;
* Previous hematopoietic stem cell transplantation;Patients can have had prior relapsed disease as long as they have never been previously transplanted;
* Known history of HIV infection;
* Use of corticosteroids (glucocorticoids) within 21 days of bone marrow collection;
* Use of any myeloma-specific therapy within 21 days of bone marrow collection;
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents within seven days of registration;
* Participation in any clinical trial within 28 days of registration on this trial, which involved an investigational drug or device;
* History of malignancy other than multiple myeloma within five years of registration, except adequately treated basal or squamous cell skin cancer;
* Active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosis) requiring active systemic treatment. Hypothyroidism without evidence of Grave's disease or Hashimoto's thyroiditis is permitted.
* Human T-lymphotropic virus (HTLV) 1 or 2 positive;
* Known hypersensitivity to Prevnar or any of its components;
* Contraindication to phosphodiesterase-5 inhibitors (e.g. currently on nitrates).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Imus, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at four sites: Johns Hopkins University, Moffitt Cancer Center, Mayo Clinic (Jacksonville) and the Blood and Marrow Transplant Group of Georgia (Northside).
Pre-assignment Details: Of the 102 patients randomized, one was randomized to the control group who was lost to follow-up prior to start; did not have aMILs harvested, and was not transplanted. This patient is therefore not included in this report.
Period: Overall Study
Arm/Group | aMIL Arm | No aMIL
Started | 70 | 31
Completed | 61 | 29
Not Completed | 9 | 2
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Disease progression | 3 | 1
Not completed — Product contamination | 2 | 0
Not completed — Failed expansion of cell product | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | aMIL Arm | No aMIL | Total
Number analyzed (Participants) | 70 | 31 | 101
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.5 [35.0 to 74.8] | 59.0 [37.1 to 75.9] | 61.7 [35.0 to 75.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 15 | 51
  Male | 34 | 16 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 14 | 8 | 22
  Other | 2 | 1 | 3
  White | 53 | 21 | 74
Region of Enrollment [Number; unit: participants]
  United States | 70 | 31 | 101
Disease Status [Count of Participants; unit: Participants]
  Newly Diagnosed | 60 | 26 | 86
  Relapsed | 10 | 5 | 15
Myeloma Prognostic Risk Signature (MYPRS) Risk Category [Count of Participants; unit: Participants] — The Myeloma Prognostic Risk Signature (MyPRS®) (Signal Genetics™) is used to estimate the underlying activity of disease progression in patients diagnosed with active multiple myeloma.
  Participants
    High Risk | 12 | 4 | 16
    Low Risk | 25 | 15 | 40
    N/A | 8 | 2 | 10
    Indeterminate | 25 | 10 | 35
70-gene expression Prognostic Risk Score (GEP-70) [Count of Participants; unit: Participants] — The 70-gene Prognostic Risk Score (GEP-70) quantifies the expression of 70 genes commonly altered in multiple myeloma. Primarily prognostic, GEP-70 assesses risk of disease relapse and survival outcomes and is the randomization stratification of the MYPRS multiple myeloma specific gene expression profile risk categories.
  Participants
    Not High Risk | 58 | 27 | 85
    High Risk | 12 | 4 | 16
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Scoring System
  0= Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self care. Totally confined to bed or chair
  5. Dead
  Participants
    0 | 27 | 7 | 34
    1 or 2 | 34 | 21 | 55
    Missing | 9 | 3 | 12
International Staging System (ISS) Multiple Myeloma Classification [Count of Participants; unit: Participants] — Prognosticates the severity of multiple myeloma and patient survival based on routinely obtained lab values.
  Stage I= Serum β2 microglobulin < 3.5 mg/l; serum albumin ≥ 3.5 g/dl; standard-risk chromosomal abnormalities (CA) and normal lactate dehydrogenase (LDH) Stage II= not stage I or Stage III Stage III= Serum β2 microglobulin ≥ 5.5 mg/L and either high-risk CA by florescent in situ hybridization (FISH) or high LDH
  Participants
    Stage I | 20 | 10 | 30
    Stage II | 19 | 7 | 26
    Stage III | 17 | 8 | 25
    missing | 14 | 6 | 20
Salmon Stage multiple myeloma classification [Count of Participants; unit: Participants] — demonstrates the correlation between the amount of myeloma and the damage it has caused based on number of bone lesions, anemia, serum calcium levels, and serum and urine light chain levels, and can be measured as myeloma cell mass (myeloma cells in billions/m2)* .
  Stage I= low cell mass (600 billion) Stage II= intermediate cell mass (600-1200 billion) Stage III= high cell mass (>1200 billion)
  Subcategory:
  A = normal renal function. B= abnormal renal function
  Participants
    IA-IB | 9 | 0 | 9
    IIA-IIB | 14 | 7 | 21
    IIIA-IIIB | 35 | 21 | 56
    missing | 12 | 3 | 15
Number of Prior Multiple Myeloma Treatments [Median (Inter-Quartile Range); unit: prior treatments] | 1 [1 to 6] | 2 [1 to 5] | 1 [1 to 6]
Time to Diagnosis [Median (Inter-Quartile Range); unit: years] | 0.53 [0.07 to 8.15] | 0.76 [0.38 to 4.80] | 0.55 [0.07 to 8.15]
Time to stem cell transplant (SCT) [Median (Inter-Quartile Range); unit: Days] | 63.0 [35.0 to 403.0] | 56.0 [33.0 to 246.0] | 60.0 [33.0 to 403.0]

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of MILs as Assessed by the Ability to Harvest, Expand, and Infuse the MILs Product
Description: Feasibility is defined as the ability to harvest, expand, and infuse the MILs product within 120 days. After treating 60 patients with MILs, we will declare MILs not feasible if we can only harvest, expand, and deliver MILs to 40 or fewer patients.
Time Frame: 120 days
Population: 71 patients were evaluable in the feasibility set: 70 randomized to the aMILs Arm, plus one patient who was not randomized due to harvest failure.
Measure: Count of Participants; unit: Participants
Arm/Group | aMIL Arm
Number analyzed (Participants) | 71
Participants
  Total number who received aMILS | 71
  Feasible | 46
  Reason not feasible- failed harvest | 1
  Reason not feasible- disease progression | 4
  Reason not feasible- death | 1
  Reason not feasible- lost to follow-up | 1
  Reason not feasible- failed expansion | 2
  Reason not feasible- cell product contamination | 2
  Reason not feasible- greater than 120 days | 14

2. Secondary Outcome: Toxicity as Determined by Total Number of Grade 3 or Higher Adverse Events
Description: Total number of adverse events grade 3 or higher that occur from MILs harvest through 60 days after transplant.
Time Frame: 60 days from aMILs harvest until day 60 after transplant
Measure: Number; unit: adverse events
Arm/Group | aMIL Arm | No aMIL
Number analyzed (Participants) | 70 | 31
adverse events | 129 | 65

3. Secondary Outcome: Overall Survival (OS)
Description: OS assessed by number of participants alive at the end of follow up period.
Time Frame: 3 years
Population: This is an analysis by intention-to-treat and only considers transplanted patients randomized to the aMILs arm.
Measure: Count of Participants; unit: Participants
Arm/Group | aMIL Arm
Number analyzed (Participants) | 70
Participants | 55

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Median PFS time equals the time of randomization (in months) until disease progression, death from any cause, or protocol deviation due to lenalidomide dosing (above 10mg), whichever occurs first.
Time Frame: 5 years
Population: This is an analysis by intention-to-treat and only considers transplanted patients randomized to the aMILs arm.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | aMIL Arm
Number analyzed (Participants) | 70
months | 21.82 [18.53 to 41.82]

ADVERSE EVENTS:
Time Frame: 60 Days from aMILs harvest until Day 60 after transplant
Arm/Group | aMIL Arm | No aMIL
All-Cause Mortality (participants affected / at risk) | 1/70 | 1/31
Serious Adverse Events (participants affected / at risk) | 64/70 | 29/31
Other Adverse Events (participants affected / at risk) | 11/70 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | aMIL Arm (N=70) | No aMIL (N=31)
Febrile neutropenia (Blood and lymphatic system disorders) | 36 (45) | 18 (22) — Grade 3 or higher Adverse Events (AEs) from aMILs harvest to 60 days following autologous stem cell transplant (ASCT)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (2) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Device related infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Diarrhea (Gastrointestinal disorders) | 8 (8) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Enterocolitis infection (Infections and infestations) | 0 (0) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Fatigue (General disorders) | 2 (2) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
fever (General disorders) | 4 (4) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
headache (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
hypophosphatemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
hypotension (Vascular disorders) | 1 (1) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
bacteremia (Infections and infestations) | 3 (3) | 2 (2) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Kidney infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
lung infection (Infections and infestations) | 2 (2) | 2 (2) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (2) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
mucosal infection (Infections and infestations) | 11 (11) | 5 (5) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
nausea (Gastrointestinal disorders) | 1 (2) | 2 (3) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
neutrophil count decreased (Blood and lymphatic system disorders) | 7 (10) | 3 (4) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
platelet count decreased (Blood and lymphatic system disorders) | 3 (7) | 4 (4) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Scrotal Infection (Infections and infestations) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Sepsis (Infections and infestations) | 2 (2) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
Stroke (Nervous system disorders) | 0 (0) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
syncope (Nervous system disorders) | 2 (2) | 2 (2) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) — Grade 3 or higher AEs from aMILs harvest to 60 days following ASCT
white blood cell decreased (Blood and lymphatic system disorders) | 2 (4) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | aMIL Arm (N=70) | No aMIL (N=31)
manufacture failure (Product Issues) | 2 (2) | 0 (0)
product contamination (Product Issues) | 1 (1) | 0 (0)
infusion related reaction (General disorders) | 8/63 (8) | 0 (0) — 63 participants in the aMILs Arm had infusions, of those, 8 had record of infusion reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT01858558/Prot_SAP_001.pdf